CLINICAL TRIAL: NCT04198727
Title: Study of the Impact of DPD Activity on the Efficacy of Capecitabine
Acronym: DPDMAX
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Collaborators: Cerbaliance (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017/15
Record Dates: First submitted 2019-12-10; First posted 2019-12-13 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Breast Neoplasm Malignant Female
MeSH Terms: interventions — Immunophenotyping; Capecitabine

STUDY DESIGN:
Intervention Model Description: This is an open-label multi-center prospective cohort study to compare the response of patients with high phenotype to patients with normal phenotype. The analyzes performed will focus on clinical and biological criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DPD activity (Experimental)
  Interventions: Other: DPD activity assessment; Drug: Capecitabine

INTERVENTIONS:
Other: DPD activity assessment — Phenotyping DPD with enzyme activity measure and uracil dosage
  Other Names: Phenotyping
Drug: Capecitabine — Capecitabine assignement at 1000mg per square meter twice daily, cycle of 21 days, 14 days of intake, 7 days of

SUMMARY:
This study evaluates the Impact of DihydroPyrimidine Dehydrogenase (DPD) activity on the efficacy of Capecitabine in patients with metastatic breast cancer. The DPD phenotype before the initiation of treatment will be assess and then the patient will be follow up during the treatment with Capecitabine up to 24 month.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18,
* Performance status 0 to 2,
* Patients with metastatic HER2 negative breast cancer,
* Patients eligible for capecitabine monotherapy at a dose of 2000 mg / m² / day, 14 days every 21 days,
* Determination of Uracil level performed according to national recommendations,
* Patients with at least one lesion evaluable according to the RECIST criteria 1.1, or presenting at least 1 hypermetabolic lesion on PET-TDM according to PERCIST 1.0 criteria. In the case of single cutaneous metastasis (s), it is required to make photographs of lesions with a measure of the lesions using a ruler,
* Patients receiving social coverage.

Exclusion Criteria:

* Performance status> 2,
* Contraindication to capecitabine monotherapy at a dose of 2000 mg / m² / day, 14 days every 21 days,
* Presence of untreated or uncontrolled symptomatic cerebral or leptomeningeal metastases (unstable corticosteroid requirements) and / or non-clinically stable in the 3 months prior to inclusion,
* History of cancer, with the exception of cancers in complete remission for more than 5 years, totally resected cutaneous basal cell carcinoma, in situ carcinoma or in situ cervical epithelioma treated,
* Vulnerable people

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
6 months objective response rate | 6 months
  The primary endpoint will be the 6-month objective response to treatment measured using the RECIST 1.1 scale, or PERCIST 1.0. The objective response is defined as the aggregation of the complete + partial response against stabilization + progression.
  The distribution of the objective response rate with respect to the value of individual lymphocyte DPD activity before treatment will be examined. This analysis will consist in comparing the objective response rate between patients with a proficient DPD phenotype, measured by lymphocyte DPD activity (> at the 3rd quartile, ie 25% of the initial population) and non-deficient patients with DPD (including phenotype). between the 13th and 75th percentiles of the initial population).

SECONDARY OUTCOMES:
6 months objective response in proficient DPD phenotype | 6 months
  RECIST 1.1 or PERCIST 1.0 criteria
Correlation between the level of lymphocyte DPD activity and uracil dosage | 1 month
Progression-free survival | 24 months
Capecitabine Toxicity using CTCAE v 5.0 | 24 months

CONTACTS AND LOCATIONS:
Locations (5):
- France (4):
  - Clinique Saint Jean, Cagnes-sur-Mer
  - Centre Azuréen de Cancérologie, Mougins
  - Clinique St Georges, Nice
  - Centre Antoine Lacassagne, Nice
- Hôpital Princesse Grâce, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No